CLINICAL TRIAL: NCT01836510
Title: Selection of Potential Predictors of Worsening Heart Failure
Acronym: BioDetectHFIV
Status: Completed | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: TA100
Record Dates: First submitted 2013-03-19; First posted 2013-04-22 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2017-05

CONDITIONS: Heart Failure
Keywords: Heart Failure; Remote Monitoring; Lung Edema; Patient Monitoring; Prediction
MeSH Terms: conditions — Heart Failure; Pulmonary Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Multicentre study with the objective to correlate heart failure hospitalizations and deaths with Home Monitoring data in ICD/CRT-D recipients, in order to identify the combination of Home Monitoring data with the greatest sensitivity and specificity in predicting Heart Failure events.

All data are prospectively collected.

DETAILED DESCRIPTION:
Home Monitoring remotely provides continuous trends of potential HF-related variables with a sampling interval of 24 hours. Although the predictive value of individual variables may be limited, a proper combination of more variables and their 24-hour sampling may allow developing a HM diagnostic algorithm to accurately predict HF worsening within given time windows.

The objective of this Study is to select the predictive variables which are most likely to be effectively included in a future algorithm.

This is a multicentre, exploratory Study with the objective to prospectively collect follow-up and Home Monitoring data from a population of subjects with indication for ICD and/or CRT-D implantation, to document HF hospitalizations and deaths and to correlate these events with HM data to identify the combination of HM data with the greatest sensitivity and specificity in predicting HF events.

Fifty first hospitalizations for worsening HF (adjudicated by an independent board) are necessary to reach the study objective (Event driven study), which were initially assumed to be generated by 650 patients fulfilling inclusion and exclusion criteria. Sample size estimation has been reviewed after an interim analysis.

ELIGIBILITY:
Inclusion Criteria:

* Left Ventricular Ejection Fraction (LVEF) ≤ 35%
* NYHA Class II or III Heart Failure
* Men and women 18 years of age or older
* Understand the nature of the procedure
* Give written informed consent

Exclusion Criteria:

* No indication or contraindication for ICD or CRT-D therapy
* Permanent AF
* NYHA Class IV Heart Failure
* Subjects with irreversible brain damage from preexisting cerebral disease;
* Subjects with acutely decompensated heart failure
* Expected heart transplantation within next six months or planned cardiac surgery within next 3 months
* Have a life expectancy of less than six months
* Presence of any disease, other than the subject's cardiac disease associated with a reduced likelihood of survival for the duration of the trial, (e.g. cancer)
* Unstable geographical residence (unable to anticipate to be resident in the area of the referring participating centre during the study period) and/or GSM-free residence
* Subjects who were not been implanted with ICD or CRT-D devices compatible with HM transmissions
* Age <18 years
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population of subjects with an indication for ICD and/or CRT-D implantation according to current guidelines
Sampling Method: Non-Probability Sample
Enrollment: 922 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
First Hospitalization for worsening Heart Failure (HF) | Participants will be followed for the duration of follow-up, an expected average of 2 years
  Hospitalization is defined as a non-elective hospital admission for medical or surgical therapy that results in at least one overnight stay.
  Hospitalization for worsening HF is defined as a hospitalization fulfilling the following criteria:
  1. It was triggered by increased symptom(s) and sign(s) OR objective evidence of worsening HF (LVEF, ECG, or other instrumental evidences);
  2. It required administration or augmentation of intravenous or oral HF medication;

SECONDARY OUTCOMES:
A composite of death for worsening heart failure, hospitalizations for worsening HF and acute interventions for worsening HF. | Participants will be followed for the duration of follow-up, an expected average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Antonio D'Onofrio, MD, Principal Investigator — A. O. dei Colli, Vincenzo Monaldi Hospital, Naples; Luigi Padeletti, Prof., Study Chair — IRCSS Multimedica, Milano
Locations (34):
- Italy (32):
  - Cliniche Humanitas Gavazzeni, Bergamo
  - Spedali Civili, Brescia
  - Di Summa Hospital, Brindisi
  - Fondazione Giovanni Paolo II, Campobasso
  - Francesco Ferrari Hospital, Casarano
  - Ospedale Sant'Anna e San Sebastiano, Caserta
  - A.O.U. Policlinico Vittorio Emanuele, Catania
  - Ospedale Bufalini, Cesena
  - Sant'Anna Hospital, Como
  - S. Croce Hospital, Cuneo
  - San Giuseppe, Empoli
  - A.O.U. Careggi, Florence
  - Mater Salutis Hospital, Legnago
  - Casa di Cura Montevergine, Mercogliano (AV)
  - Azienda Ospedaliera Ospedali Riuniti Papardo Piemonte, Messina
  - A. O. Monaldi, Naples
  - Policlinico Federico II, Napoli
  - ARNAS Civico, Palermo
  - S. Maria della Misericordia, Perugia
  - Ospedale Civile, Piacenza
  - S. Maria degli Angeli Hospital, Pordenone
  - Ospedale San Pietro, Rome
  - Policlinico Casilino, Rome
  - San Filippo Neri, Rome
  - A.O.U. San Giovanni di Dio Ruggi d'Aragona, Salerno
  - IRCCS Multimedica, Sesto San Giovanni
  - Santissima Annunziata Hospital, Taranto
  - S. Maria di Ca' Foncello Hospital, Treviso
  - A.O.U. Ospedali Riuniti, Trieste
  - Ospedale di Circolo e Fondazione Macchi, O.U. Cardiology II, Varese
  - Ospedale di Circolo e Fondazione Macchi, O.U. Cardiology I, Varese
  - Guzzardi Hospital, Vittoria (RG)
- Spain (2):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario Virgen de la Victoria, Málaga

REFERENCES:
- [Derived] Padeletti L, Botto GL, Curnis A, De Ruvo E, D'Onofrio A, Gronda E, Ricci RP, Vado A, Zanotto G, Zecchin M, Antoniou X, Gargaro A. Selection of potential predictors of worsening heart failure: rational and design of the SELENE HF study. J Cardiovasc Med (Hagerstown). 2015 Nov;16(11):782-9. doi: 10.2459/JCM.0000000000000171. PMID 25036269